CLINICAL TRIAL: NCT06124638
Title: Clinical Evaluation of the Panbio™ COVID-19/Flu A&B Panel to Support Home Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2324101
Record Dates: First submitted 2023-11-08; First posted 2023-11-09 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Influenza A; Influenza Type B
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-Testing Group (Experimental): Lay users (self-tester or caregiver) will be provided with a Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test kit. Each lay user will collect one mid-turbinate nasal swab from both nostrils, perform and interpret the Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test. All procedures for testing and result interpretation, including sample collection and extraction will be conducted by the lay user following the Instructions for Use provided in the kit. Participants will be asked to document their result interpretation and will pass the test to site staff, who will document their interpretation of the result. In addition, a second swab will be collected by study staff and eluted in Viral Transport Medium (VTM).
  Interventions: Diagnostic Test: Panbio™ COVID-19/Flu A&B Panel

INTERVENTIONS:
Diagnostic Test: Panbio™ COVID-19/Flu A&B Panel — The Panbio™ COVID-19/Flu A&B Rapid Panel Self-Test device is a visual lateral flow assay, for rapid immunochromatographic qualitative detection of COVID-19 antigen, Influenza A antigen and Influenza B antigen in self-collected mid-turbinate nasal swabs. The test is designed to be used by lay users.

SUMMARY:
This study is designed to demonstrate the performance and usability of the the Panbio™ COVID-19/Flu A&B Panel Self Test in the hands of patients/lay-users. Nasal swabs will be self-collected by subjects/lay-users who are symptomatic and suspected of viral respiratory infection. They will perform, read, and interpret the test result. The test is intended for nonprescription home use for qualitative detection of COVID-19, Influenza A antigen, and Influenza B antigen.

DETAILED DESCRIPTION:
The total number of anterior nasal swabs collected from each consented Participant is two (2). Participants at least two (2) years of age meeting eligibility criteria will be enrolled.

The order of nasal swab collection will be randomized according to the Participant ID as to which swab is used for Panbio™ COVID-19/Flu A&B Panel Self Test and which is to be eluted into VTM for comparator testing. Site staff should allow for a minimum 15 minute period between the 2 swabs to allow for normalization of the swabbing site. For Participants with an odd numbered Participant ID, the first swab collected will be used for Panbio™ COVID-19/Flu A&B Panel Self Test and the second swab collected will be eluted into VTM for comparator testing. For Participants with an even numbered Participant ID, the first swab collected will be eluted into VTM for comparator testing and the second swab collected will be used for Panbio™ COVID-19/Flu A&B Panel Self Test.

Sample collection for the Self Test:

Each Participant (lay user who will be a self-tester or caregiver) from whom informed consent has been obtained will be provided a single use test kit containing a Panbio™ COVID-19/Flu A&B Panel Self Test and a sterile nasal swab. The Participant will self-collect one (1) anterior nasal swab, perform the Panbio™ COVID- 19/Flu A&B Panel Self Test, then interpret and record the result. Parents of pediatric participants under the age of 14 or Legally Authorized Representatives of adult Participants unable to perform self-collection will collect one (1) anterior nasal swab from the Participant, perform the Panbio™ COVID-19/Flu A&B Panel Self Test, then interpret and record the result. To simulate a home environment testing will occur in a designated room/area that does not contain medical equipment. The designated room/area will at minimum contain a table/counter, chair and lamp for testing. The participant will be provided with the Instructions for Use prior to testing. Participants will not be able to observe other participants conducting testing. The Participant will follow Panbio instructions to insert the swab up to one inch first into the right nostril, to rotate/swirl the swab five (5) times to obtain sample, then remove and insert the same swab into the left nostril, repeating the rotate/swirl technique. After sample collection, Participants will test the sample on the Panbio™ COVID-19/Flu A&B Panel Self Test and interpret the results. Participants will be asked to document their result interpretation, and will pass the completed test to site staff, who will independently and separately document their interpretation of the result. Site staff will interpret the test immediately and at the same time photograph the test result. Site staff will be blinded to the test result recorded by the Participant. Participants/lay users, caregivers, and site staff will be blinded to a Participant's standard of care COVID-19 and/or Flu test results.

Sample collection for the comparator:

Site staff will collect one (1) anterior nasal swab from the Participant by inserting the swab 1-2 cm into one of the anterior nares. Staff will rotate the swab against the nasal mucosa for about 3 seconds and withdraw. Staff will repeat with the other anterior nare using the same swab, and vigorously elute the swab in Viral Transport Medium (VTM). VTM will be send to the central lab and be tested with reverse transcriptase - Polymerase Chain Reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least two (2) years of age, and
* Participant is suspected of acute viral respiratory infection by a healthcare professional, and
* Participant is within seven (7) days of symptom onset, and
* Participant is experiencing two or more of the following symptoms

  * Fever of >100.0°F/ 37.8°C
  * Cough
  * Fatigue
  * New loss of taste or smell
  * Congestion or runny nose
  * Shortness of breath or difficulty breathing
  * Sore throat
  * Muscle or body aches
  * Headache
  * Nausea or vomiting
  * Diarrhea

Exclusion Criteria:

* Participant is currently enrolled in a study to evaluate an investigational drug or experimental treatment
* Participants with an active nosebleed
* Participant has undergone a nasal wash or nasal aspirate procedure on day of enrolment
* Participant has received a nasal spray or mist Influenza vaccine (i.e. FluMist) within the last 30 days
* Participant has tested positive for COVID-19 within the last 45 days (excluding test results received after current onset of symptoms)
* Participant has received antiviral medications for Influenza (Amantadine, Rimantadine, Ribavirin, Oseltamivir, Zanamivir) in the previous 45 days
* Participant has received medication or treatment for COVID-19 infection in the last 45 days (including antivirals, convalescent plasma therapy, monoclonal antibody treatment (mAb), Remdesivir, long-acting antibody (LAAB) treatment (Evusheld)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the Panbio™ COVID-19/Flu A&B Rapid Panel device | 6 months
  The primary objective of this study is to demonstrate the positive and negative percent agreement (PPA and NPA) of the Panbio™ COVID-19/Flu A&B Panel Self Test against the comparator Roche cobas® SARS-CoV-2 (K231306) and Quidel Lyra® Influenza A+B Assay (K230236), in symptomatic patients suspected of respiratory viral infection, when nasal swabs are self-collected by the patient/lay user. The patient/lay user will perform the test, read and interpret the test result.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cahaba Research Inc, Pelham, Alabama
  - Maimonides Medical Center, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No